CLINICAL TRIAL: NCT06854315
Title: Effect of a ChatGPT-Based Digital Counseling Intervention on Anxiety and Depression in Patients With Cancer: A Prospective, Randomized Trial
Brief Title: Effect of ChatGPT-Based Digital Counseling on Anxiety and Depression in Cancer: A Randomized Trial
Acronym: ONCO-AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Orhun Akdoğan, Medical Oncologist, Gazi University Faculty of Medicine, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-1096068; E-1096068 (Other: Gazi University Faculty of Medicine)
Record Dates: First submitted 2025-02-19; First posted 2025-03-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Anxiety; Depression; Artifical Intelligence
Keywords: Artificial Intelligence; Cancer Patient Education; Supportive Care; AI-Based Counseling
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model in which participants were randomly assigned to one of two groups: (1) the ChatGPT-assisted counseling group, which received standard chemotherapy education plus access to ChatGPT for personalized inquiries, or (2) the control group, which received standard clinician-led chemotherapy education alone. Both groups were followed simultaneously to assess changes in anxiety and depression levels before the second chemotherapy cycle.
Who Masked: Outcomes Assessor
Masking Description: This study used an outcomes assessor-blinded design, meaning that the researchers responsible for analyzing the primary and secondary outcomes were blinded to group allocation. However, participants, care providers, and investigators were aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ChatGPT-Arm (Experimental): Participants in this group received standard clinician-led chemotherapy education plus access to ChatGPT-based digital counseling. They were allowed to submit up to 10 personalized questions to ChatGPT regarding their treatment. All AI-generated responses were reviewed for accuracy by oncology specialists.
  Interventions: Behavioral: ChatGPT-Based Digital Counseling
- Control Group (Other): Standard pre-chemotherapy education was provided by oncologists and oncology nurses, covering expected side effects, treatment protocols, and general supportive care.
  Interventions: Behavioral: Standard Clinician-Led Education

INTERVENTIONS:
Behavioral: ChatGPT-Based Digital Counseling — Participants in this group received standard clinician-led chemotherapy education plus access to ChatGPT-based digital counseling. They could submit up to 10 personalized questions regarding their treatment, side effects, and supportive care. Oncology specialists reviewed ChatGPT-generated responses for accuracy. This intervention aimed to assess whether AI-assisted counseling could reduce anxiety and depression levels in newly diagnosed cancer patients.
  Arms: ChatGPT-Arm
Behavioral: Standard Clinician-Led Education — Participants in this group received only standard clinician-led chemotherapy education, delivered by oncology physicians and nurses. The education covered key aspects of chemotherapy, including potential side effects, treatment schedules, and supportive care recommendations. Unlike the ChatGPT group, these participants did not receive AI-assisted counseling or additional interactive educational tools.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the impact of a ChatGPT-based digital counseling intervention on anxiety and depression in newly diagnosed cancer patients undergoing chemotherapy. Patients are randomly assigned to one of two groups:

ChatGPT Group: Patients receive standard chemotherapy education plus access to ChatGPT, where they can ask up to 10 personalized questions about their treatment.

Control Group: Patients receive only standard chemotherapy education provided by oncologists and nurses.

The primary outcome is the change in anxiety and depression levels, measured using the Hospital Anxiety and Depression Scale (HADS), recorded at baseline and before the second chemotherapy cycle.

Secondary outcomes include patient engagement patterns, the types of questions asked, and an assessment of ChatGPT's responses by oncologists.

This study seeks to explore whether AI-based digital counseling can serve as a complementary support tool for newly diagnosed cancer patients.

DETAILED DESCRIPTION:
Study Design This prospective, randomized controlled trial aims to evaluate the effects of a ChatGPT-based digital counseling intervention on anxiety and depression in newly diagnosed cancer patients undergoing chemotherapy.

The study is conducted at two oncology centers between July 2024 and December 2024. Patients are randomly assigned (1:1) to either:

ChatGPT-Assisted Counseling Arm: Patients receive standard chemotherapy education plus the ability to ask up to 10 personalized questions to ChatGPT. All AI-generated responses are reviewed for accuracy by oncology specialists.

Standard Education Arm: Patients receive only clinician-led chemotherapy education, without AI-based support.

Primary and Secondary Outcomes

Primary Outcome: Change in Hospital Anxiety and Depression Scale (HADS-A, HADS-D) scores between baseline and prior to the second chemotherapy cycle.

Secondary Outcomes:

Differences in patient engagement behaviors and information-seeking patterns. Analysis of the accuracy and reliability of ChatGPT-generated responses. The role of AI in addressing sensitive or under-discussed topics in oncology education (e.g., sexual health, alternative medicine).

Statistical Analysis The sample size is estimated based on detecting a 2-point difference in HADS scores (α=0.05, power=80%).

Nonparametric tests (Mann-Whitney U test, Wilcoxon signed-rank test) are planned for within- and between-group comparisons.

Multivariable logistic regression will assess independent predictors of anxiety reduction.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years Newly diagnosed solid tumor (treatment-naïve) Scheduled to begin first-line chemotherapy ECOG performance status ≤2 Sufficient cognitive function to understand and complete the Hospital Anxiety and Depression Scale (HADS) questionnaire Ability to provide written informed consent

Exclusion Criteria:

Recurrent or metastatic cancer requiring urgent treatment Cognitive impairment that affects the ability to understand or complete the Hospital Anxiety and Depression Scale (HADS) questionnaire Severe psychiatric disorders (e.g., schizophrenia, bipolar disorder, severe major depressive disorder) that could interfere with study participation Concurrent participation in another interventional study related to psychological support or digital counseling

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety and Depression Scores (HADS-A and HADS-D) | Time Frame: Change in Hospital Anxiety and Depression Scale (HADS-A, HADS-D) scores from baseline to prior to the second chemotherapy cycle (each cycle is 21 days).
  The primary outcome is the change in Hospital Anxiety and Depression Scale (HADS-A, HADS-D) scores between baseline and the second chemotherapy cycle. The difference between groups will be assessed to determine the impact of ChatGPT-assisted counseling on anxiety and depression levels in newly diagnosed cancer patients.

SECONDARY OUTCOMES:
Differences in Patient Engagement and Information-Seeking Behavior | Change in Hospital Anxiety and Depression Scale (HADS-A, HADS-D) scores from baseline to prior to the second chemotherapy cycle (each cycle is 21 days).
  The number and type of questions asked by participants in the ChatGPT-assisted group will be analyzed to assess differences in information-seeking behavior compared to the standard education group.
Accuracy and Reliability of ChatGPT Responses | Baseline and Day 21 (prior to Cycle 2, each cycle is 21 days)
  The oncology specialists will review all AI-generated responses and classify them as "appropriate," "inappropriate," or "unreliable." The percentage of correct responses will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara, Yenimahalle
  - Gazi University Faculty of Medicine, Department of Medical Oncology, Ankara, Yenimahalle

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and institutional policies. The dataset contains sensitive patient information, and sharing is not planned to ensure patient confidentiality and compliance with ethical guidelines.

REFERENCES:
- [Background] Akdogan O, Uyar GC, Yesilbas E, Baskurt K, Malkoc NA, Ozdemir N, Yazici O, Oksuzoglu B, Uner A, Ozet A, Sutcuoglu O. Effect of a ChatGPT-based digital counseling intervention on anxiety and depression in patients with cancer: A prospective, randomized trial. Eur J Cancer. 2025 May 15;221:115408. doi: 10.1016/j.ejca.2025.115408. Epub 2025 Apr 3. PMID 40215593